CLINICAL TRIAL: NCT04340401
Title: A Phase II Study of Total Neoadjuvant Chmoradiation Treatment Plus SHR1210 for High-risk Locally Advanced Rectal Cancer and Biomarker Screening Base on Neoantigen
Brief Title: Total Neoadjuvant Treatment Plus SHR1210 for High-risk Rectal Cancer and Biomarker Screening Base on Neoantigen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, Chief, Unit III & Ostomy Service, Gastrointestinal Cancer center, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH-R04
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Rectal Cancer
Keywords: High-risk locally advanced Rectal cancer; SHR-1210; Total Neoadjuvant chmoradiation Treatment; pCR rate
MeSH Terms: conditions — Rectal Neoplasms | interventions — camrelizumab; Oxaliplatin; Capecitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TNT+SHR1210 (Experimental): Patients with high-risk locally advanced rectal cancer will receive chemotherapy and SHR-1210 before chemoradiaton, after chemoradiaton, patient will receive consolidation chemotherapy. This arm is called Total Neoadjuvant Treatment (TNT) plus SHR-1210. The neoadjuvant chemotherapy regimen is designed as 3 cycles of CapeOX ( Capecitabine + Oxaliplatin ) plus SHR-1210 over a period of approximately 8 weeks. Tumor response will be evaluated after chemotherapy. Then patients will undergo 22f-IMRT (Intensity modulated radiotherapy) with capecitabine. Patients will receive two more cycles of consolidation CapeOX if tolerable when there was no progressed disease in induction CapeOX.
  Finally, patients will receive TME (Total mesorectal excision) following TNT+SHR1210 if no metastasis occurs.
  Interventions: Drug: SHR-1210; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Intensity modulated radiotherapy; Procedure: Total mesorectal excision

INTERVENTIONS:
Drug: SHR-1210 — Patients will receive 3 cycles induction CapeOX and SHR-1210
  Other Names: Camrelizumab
Drug: Oxaliplatin — CapeOX is a combination chemotherapy regimen with OXA and CAPE, patients with high-risk rectal cancer will receive 3 cycles induction CapeOX and SHR-1210, intensity modulated radiotherapy with concurrent capecitabine and 2 cycles consolidation CapeOX and total mesorectal excision.
  Other Names: OXA
Drug: Capecitabine — CapeOX is a combination chemotherapy regimen with OXA and CAPE, patients with high-risk rectal cancer will receive 3 cycles induction CapeOX and SHR-1210, intensity modulated radiotherapy with concurrent capecitabine and 2 cycles consolidation CapeOX and total mesorectal excision.
  Other Names: CAPE
Radiation: Intensity modulated radiotherapy — patients will receive intensity modulated radiotherapy with capecitabine
  Other Names: IMRT
Procedure: Total mesorectal excision — Patients will receive TME (Total mesorectal excision) following TNT+SHR1210 if no metastasis occurs.
  Other Names: TME

SUMMARY:
This study is designed to test the efficacy and safety of Total Neoadjuvant Treatment plus SHR1210（an anti-PD-1 Inhibitor) for High-risk locally advanced Rectal Cancer, Meanwhile, screening effective Biomarker base on neoantigen.

DETAILED DESCRIPTION:
The combined treatment model of neoadjuvant chemoradiotherapy treatment + radical rectal resection + adjuvant therapy has become the standard treatment model for locally advanced mid-low rectal cancer, However, the existing evidence shows that this comprehensive treatment method has reached the upper limit of efficacy and cannot continue to reduce the metastatic rate and improve the survival rate.

Recent studies have shown that PD-1 antibody inhibitors have excellent curative effects on the treatment of a variety of tumors and have good safety.

This study is a single-arm, single-center, prospective, phase II clinical study. It is designed to test the efficacy and safety of Total Neoadjuvant chmoradiation Treatment plus SHR1210 for High-risk locally advanced Rectal Cancer, Meanwhile, screening effective Biomarker base on neoantigen.

In this study, patients with high-risk rectal cancer will receive 3 cycles induction CapeOX and SHR-1210, intensity modulated radiotherapy with concurrent capecitabine and 2 cycles consolidation CapeOX and total mesorectal excision.

This study is designed to recruit 25 patients in all.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤70 years.
* ECOG Performance status 0-1.
* Histologically confirmed diagnosis of adenocarcinoma of the rectum.
* The distance from down verge of tumor to anal-rectal junction (ARJ) ≤8cm, or ≤12 cm based on sigmoidoscopy.
* Clinical Stage T3c, T3d, T4a or T4b, or EMVI (+) or mrN2 or MRF (+) based on MRI.
* No evidence of distant metastases.
* No prior pelvic radiation therapy.
* No prior chemotherapy or surgery for rectal cancer.
* No active infections requiring systemic antibiotic treatment.
* No systemic infection requiring antibiotic treatment.
* No immune system disease.
* ANC > 1.5 cells/mm3, HGB > 9.0 g/dL, PLT > 100,000/mm3, total bilirubin≤ 1.5×ULN, AST≤ 2.5×ULN, ALT ≤ 2.5×ULN.
* Serum creatinine is within 1.5 times the physiological range， creatinine clearance rate≥50 ml/min
* Patients with controllable hypertension were included.
* Patients who did not receive anticoagulant therapy: INR, aPTT is required to be within the 1.5 times the physiological range;Patients who receive anticoagulant therapy: INR, aPTT is required to be within the physiological range.
* FT3, FT4, TSH are Normal or abnormal without clinical significance.
* ECG examination is Normal or abnormal without clinical significance; Echocardiography shows that LVEF>50%.
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.
* Patients show good adherence, follow -up on time. It is recommended that all patients provide tumor tissue samples (preferably fresh tissue samples) for pathological genetic testing prior to enrollment.
* Fertile men or women with potential for pregnancy must use highly effective contraception throughout the trial. And continue contraception for 12 months after treatment ends.

Exclusion Criteria:

* Recurrent rectal cancer.
* Anticipated unresectable tumor after neoadjuvant treatment.
* Patients with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer.
* Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA.
* Other Anticancer or Experimental Therapy.
* Women who are pregnant or breast-feeding.
* Patients with any other concurrent medical or psychiatric condition or disease which would make them inappropriate candidates for entry into this study.
* Patients with a history of anti-PD-1, anti-PD-L1, anti-PD-L2 or CEGFR TKI therapy.
* Patients underwent major surgery or had not recovered from the side effects of this surgery, received a vaccine, received immunotherapy within 4 weeks before the first use of the study drug, and received radiotherapy within 2 weeks.
* Patients who received hematopoietic stimulating factors therapy, such as G-CSF and erythropoietin, within 1 week before the first administration of the study drug.
* Patients are allergic to study medication and its ingredients.
* Patients have active lung disease (such as interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or active tuberculosis.
* Patients have any uncontrollable clinical problems, including but not limited to:

  1. Persistent or severe infection.
  2. Hypertension that can't be effectively controlled by drugs（ blood pressure reading of 150 over 90）.
  3. Uncontrolled diabetes
  4. Heart disease (Class III / IV congestive heart failure or cardiac block as defined by the New York Heart Association)
  5. Patient has or is suspected of having an autoimmune disease,Such as pituitary inflammation, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc.
* Patients have other serious, acute or chronic diseases or have abnormal test results, and the investigator judges that this may increase the patient's risk of participating in the trial or interfere with the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate(pCR rate) | 1 month after surgery
  The number of patients with pCR divided by the total number of patients

SECONDARY OUTCOMES:
Toxicity of TNT+SHR-1210 | 90 days after neoadjuvant treatment
  Category and grade of adverse event during neoadjuvant chemotherapy
Change of TCR repertoire | 1 week before surgery
  Use neoantigen model to find biomarkers related to the effect of TNT+SHR1210 for patients with rectal cancer; compare and analyze the differences in TCR repertoire changes in peripheral blood.
Disease-free survival (DFS) | 3 years
  The 3-year DFS will be defined as the percentage of patients alive without local recurrence or distant metastasis of disease at 3 years measured from the date of the administration of treatment.
Surgical complication rate | 30 days after surgery
  Rate of patients who had surgical complications during the perioperative period
Major adverse events | 90 days after the last use of SHR-1210
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China